CLINICAL TRIAL: NCT02485899
Title: A Multicenter, Multinational, Extension Study to Evaluate the Long-Term Efficacy and Safety of BMN 190 in Patients With CLN2 Disease
Brief Title: An Extension Study to Evaluate the Long-Term Efficacy and Safety of BMN 190 in Patients With CLN2 Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190-202
Record Dates: First submitted 2015-04-24; First posted 2015-06-30 (Estimated); Results first posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-07

CONDITIONS: Jansky-Bielschowsky Disease; Batten Disease; Late-Infantile Neuronal Ceroid Lipofuscinosis Type 2; CLN2 Disease; CLN2 Disorder
Keywords: Late infantile Neuronal Ceroid Lipofuscinosis Type 2; LINCL; NCL2; CLN2; Jansky-Bielschowsky disease
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses | interventions — cerliponase alfa

STUDY DESIGN:
Intervention Model Description: Because of practical (limited number of available patients) and ethical (neurosurgery in children with fatal neurologic disease) concerns, this study design could not involve contemporaneous, matched, randomized, blinded, or untreated control subjects. As such, data from the DEM-CHILD Multi-Center Clinical NCL Database at the University Medical Center in Hamburg, Germany (NCT04613089) was used as a control group (i.e., Natural History [NH] comparator) to determine the primary efficacy outcome measures for this study. The NH comparator was comprised of subjects from the DEM-CHILD database who satisfied the 190-201 inclusion criterion: Age ≥ 3, and at least one ML score ≥ 3 at age ≥ 3 years and further, who had at least two CLN2 assessments with values within the range 1 - 5 and at least 6 months apart.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- BMN190 recombinant human tripeptidyl peptidase-1 (rhTPP1) (Experimental): All 190-202 study subjects administered BMN 190 300 mg by continuous Intracerebroventricular (ICV) infusion at a rate of 2.5 mL/hour for approximately 4 hours) every 14 days.
  Interventions: Biological: BMN 190; Device: Intracerebroventricular (ICV) access device

INTERVENTIONS:
Biological: BMN 190 — 300 mg Intracerebroventricular (ICV) infusion administered every other week for up to 240 weeks
  Other Names: recombinant human tripeptidyl peptidase-1 (rhTPP1); cerliponase alfa
Device: Intracerebroventricular (ICV) access device — Surgical implantation of an MRI compatible ICV access device in the lateral ventricle of the right hemisphere is required for administration of study drug.

SUMMARY:
The Phase 1/2 study (190-201) evaluated the efficacy and safety of a 300 mg dose of BMN 190 administered every other week (qow) to patients with CLN2. The dose and regimen for this study (190-202) are based on the results of the 190-201 study. The rationale for this phase 2 extension study is to provide patients who complete the 190-201 study with the option to continue BMN 190 treatment. The 190-202 study is an open label extension protocol to assess long-term safety and efficacy.

DETAILED DESCRIPTION:
BMN 190 is a recombinant form of human tripeptidyl peptidase 1 (TPP1), the enzyme deficient in patients with CLN2 disease (also known as classical late-infantile CLN2, cLINCL, or Jansky-Bielschowsky disease), a form of Batten Disease. As an enzyme replacement therapy (ERT), BMN 190 is designed to help restore TPP1 enzyme activity. The Phase 1/2 study (190-201) evaluated the efficacy and safety of a 300 mg dose of BMN 190 administered every other week (qow) to patients with CLN2. The dose and regimen for this study (190-202) are based on the results of the 190-201 study. The rationale for this phase 2 extension study is to provide patients who complete the 190-201 study with the option to continue BMN 190 treatment. The 190-202 study is an open label extension protocol to assess long-term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed 48 weeks in Study 190-201.
* Is willing and able to provide written, signed informed consent. Or, in the case of patients under the age of 18 (or other age as defined by regional law or regulation), provide written assent (if required) and have written informed consent, signed by a legally authorized representative, after the nature of the study has been explained, and prior to performance of research-related procedures.
* Males and females who are of reproductive age should practice true abstinence, defined as no sexual activity, during the study and for 6 months after the study has been completed (or withdrawal from the study). If sexually active and not practicing true abstinence, males and females of reproductive age must use a highly effective method of contraception while participating in the study.
* If female, of childbearing potential, must have a negative pregnancy test at the Screening Visit and be willing to have additional pregnancy tests done during the study.

Exclusion Criteria:

* Has had a loss of 3 or more points in the combined motor and language components of the Hamburg CLN2 rating scale between Baseline of Study 190-201 and the Study Completion visit in Study 190-201 and would not benefit from enrolling in the study in the Investigator's discretion.
* Has a score of 0 points on the combined motor and language components of the Hamburg CLN2 rating scale.
* Is pregnant or breastfeeding, at Baseline, or planning to become pregnant (self or partner) at any time during the study.
* Has used any investigational product (other than BMN 190 in 190-201), or investigational medical device, within 30 days prior to Baseline; or is required to use any investigational agent prior to completion of all scheduled study assessments.
* Has a concurrent disease or condition that would interfere with study participation, or pose a safety risk, as determined by the Investigator.
* Has any condition that, in the view of the Investigator, places the patient at high risk of poor treatment compliance or of not completing the study.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — BioMarin Pharmaceutical
Locations (4):
- Nationwide Children's Hospital, Columbus, Ohio, United States
- Universitaetsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Children's Hospital Bambino Gesù,IRCCS, Rome, Piazza, Italy
- Great Ormond Street Childrens Hospital, London, United Kingdom

REFERENCES:
- [Derived] Specchio N, Gissen P, de Los Reyes E, Olaye A, Camp C, Curteis T, Griffiths A, Butt T, Cohen-Pfeffer J, Slasor P, Sisic Z, Jain M, Schulz A. Exploring concurrent validity of the CLN2 Clinical Rating Scale: Comparison to PedsQL using cerliponase alfa clinical trial data. PLoS One. 2024 May 22;19(5):e0302382. doi: 10.1371/journal.pone.0302382. eCollection 2024. PMID 38776275
- [Derived] Schulz A, Specchio N, de Los Reyes E, Gissen P, Nickel M, Trivisano M, Aylward SC, Chakrapani A, Schwering C, Wibbeler E, Westermann LM, Ballon DJ, Dyke JP, Cherukuri A, Bondade S, Slasor P, Cohen Pfeffer J. Safety and efficacy of cerliponase alfa in children with neuronal ceroid lipofuscinosis type 2 (CLN2 disease): an open-label extension study. Lancet Neurol. 2024 Jan;23(1):60-70. doi: 10.1016/S1474-4422(23)00384-8. PMID 38101904
- [Derived] Gissen P, Specchio N, Olaye A, Jain M, Butt T, Ghosh W, Ruban-Fell B, Griffiths A, Camp C, Sisic Z, Schwering C, Wibbeler E, Trivisano M, Lee L, Nickel M, Mortensen A, Schulz A. Investigating health-related quality of life in rare diseases: a case study in utility value determination for patients with CLN2 disease (neuronal ceroid lipofuscinosis type 2). Orphanet J Rare Dis. 2021 May 12;16(1):217. doi: 10.1186/s13023-021-01829-x. PMID 33980287
- [Derived] Schulz A, Ajayi T, Specchio N, de Los Reyes E, Gissen P, Ballon D, Dyke JP, Cahan H, Slasor P, Jacoby D, Kohlschutter A; CLN2 Study Group. Study of Intraventricular Cerliponase Alfa for CLN2 Disease. N Engl J Med. 2018 May 17;378(20):1898-1907. doi: 10.1056/NEJMoa1712649. Epub 2018 Apr 24. PMID 29688815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 190-201 was conducted at 5 clinic sites in Germany, Italy, the United Kingdom and the United States. One subject from one of the two 190-201 sites in the United Kingdom withdrew after 1 dose of BMN 190 and therefore this site was not activated in 190-202.
  The comparator group for determination of the primary efficacy outcome measures in this study was comprised of 42 Natural History (NH) subjects with CLN2 disease selected from the DEM-CHILD database (NCT04613089).
Pre-assignment Details: 190-202 is the extension of treatment & follow-up for subjects enrolled in Study 190-201. The ITT analysis population was comprised of the 23 subjects who completed the 190-201 study and enrolled in the 190-202 study (completed 48 weeks in 190-201, met all other 190-202 study inclusion criteria and to whom none of the 190-202 study exclusion criteria applied). The safety analysis population in Study 190-202 was comprised of the 24 subjects in Study 190-201 who had an ICV access device implanted.
Groups:
- 190-202 (300 mg): 190-202 Intent to Treat (ITT)/Efficacy Population (n = 23): The 23 subjects who completed the 190-201 study and enrolled in the 190-202 study (i.e., completed 48 weeks in Study 190-201, met all other 190-202 study inclusion criteria and to whom none of the 190-202 study exclusion criteria applied).
  190-202 Safety Population (n = 24): All study subjects who had an ICV access device implanted in Study 190-201.
- Natural History Comparator: The NH comparator population consisted of subjects from the DEM-CHILD database who satisfied the 190-201 inclusion criterion: Age ≥ 3 years; and at least one ML score ≥3 points at age ≥3 years and further, who had at least two CLN2 assessments with values within the range 1 to 5 points and at least 6 months apart.
Period: Overall Study
Arm/Group | 190-202 (300 mg) | Natural History Comparator
Started | 24 | 42 (The control group (NH comparator) used for determination of the primary efficacy outcomes of this study was comprised of data from 42 subjects with CLN2 disease from the DEM-CHILD database (NCT04613089).)
Completed | 17 | 42 (The control group (NH comparator) used for determination of the primary efficacy outcomes of this study was comprised of data from 42 subjects with CLN2 disease from the DEM-CHILD database (NCT04613089).)
Not Completed | 7 | 0
Not completed — Protocol-Specified Withdrawal Criterion Met | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal by Parent/ Guardian | 4 | 0

BASELINE CHARACTERISTICS:
Population: The demographic characteristics of the enrolled population are summarized for the 190-201/202 study (24 subjects). The demographic characteristics of the control group (NH comparator) which were necessary to determine the primary efficacy outcome measures, are also included (42 subjects).
Groups:
- Natural History Comparator: Because of practical (limited number of available patients) and ethical (neurosurgery in children with fatal neurologic disease) concerns, this study design could not involve contemporaneous, matched, randomized, blinded, or untreated control subjects. As such, data from the DEM-CHILD Multi-Center Clinical NCL Database at the University Medical Center in Hamburg, Germany (NCT04613089) was used as a control group (i.e., Natural History [NH] comparator) to determine the primary efficacy outcome measures for this study. The control group (NH comparator) was comprised of subjects from the DEM-CHILD database who satisfied the 190-201 inclusion criterion: Age ≥ 3, and at least one ML score ≥ 3 at age ≥ 3 years and further, who had at least two CLN2 assessments with values within the range 1 - 5 and at least 6 months apart.
- Total: Total of all reporting groups
Arm/Group | 190-202 (300 mg) | Natural History Comparator | Total
Number analyzed (Participants) | 24 | 42 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] — Age immediately preceding the first 300 mg infusion.
  Data for Study 190-201, was recorded as the number of complete (integer) years lived at the time of study enrollment. Data presented for 190-201/202 is based on derived age (continuous variable) using the baseline date compared to the date of birth considering both month and year of birth.
  The change from reporting "age at enrollment" for 190-201 to reporting "age at baseline" for 190-201/202 was made to align with the reported outcome measure of baseline ML score.
  years | 5.0 (1.29) | 4.0 (0.92) | 4.3 (1.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 9 | 25 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 0 | 23
  Unknown or Not Reported | 0 | 42 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 23 | 0 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 42 | 42
300 mg Baseline ML Score [Mean (Standard Deviation); unit: units on a scale] — The combined motor/gait and language (ML) score, as derived from the Hamburg CLN2 rating scale, immediately preceding the first 300 mg infusion. The combined ML score is determined as the sum of the 0-3 point motor (M) and language (L) subscales where 0 represents no function, and 3 represents normal function, and can range from 0 (severely impaired) to 6 (normal).
  units on a scale | 3.5 (1.18) | 4.5 (0.77) | 4.1 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Probability of Unreversed 2-point Decline in Motor-language (ML) Score or Score of 0
Description: Motor and Language are each 0-3 point subscales in which 3 represents best function and 0 represents loss of function. Thus, the 0-6 point ML score was used as the primary mode of evaluation of loss of function.
  In 190-201, the primary endpoint was a responder endpoint: unreversed ML 2-point decline or score of 0 at Week 48 compared to the 50% rate expected in natural history using the 1-sample binomial test. For 190-202, the primary endpoint was revised to assess response over the full duration of follow-up. It is not clear, given the variable follow-up much greater than 48 weeks, what response rate is expected in natural history. For this reason, the assessment of the primary endpoint is based on comparing to natural history data and using the Kaplan-Meier method and Cox proportional hazards model with covariate adjustment (i.e., baseline ML score and age as continuous covariates, and genotype [common alleles] and sex as categorical covariates).
Time Frame: Up to Week 289
Population: BMN 190-202: 24 subjects were enrolled in 190-201 at 5 clinic sites worldwide. One subject terminated from 190-201 after a single infusion and is not included in the Intent-to-Treat (ITT) population for 190-202. Study 190-202 final efficacy results include pooled data from the complete dataset from Study 190-201 & Study 190-202 for all subjects who received >1 dose (N=23).
  NH: 42 subjects from DEM-CHILD database satisfying the criteria listed in the Arm/Group description below.
Measure: Number (95% Confidence Interval); unit: Probability of decline
Groups:
- BMN 190-202 (300 mg): All study subjects administered BMN 190 300 mg by continuous Intracerebroventricular (ICV) infusion at a rate of 2.5 mL/hour for approximately 4 hours) every 14 days.
- Natural History Comparator: The control group (NH comparator) was comprised of subjects from the DEM-CHILD database who satisfied the 190-201 inclusion criterion: Age ≥ 3, and at least one ML score ≥ 3 at age ≥ 3 years and further, who had at least two CLN2 assessments with values within the range 1 - 5 and at least 6 months apart.
Arm/Group | BMN 190-202 (300 mg) | Natural History Comparator
Number analyzed (Participants) | 23 | 42
Probability of decline
  Probability of decline: Week 49 | 0.13 [0.04 to 0.35] | 0.48 [0.34 to 0.64]
  Probability of decline: Week 97 | 0.22 [0.10 to 0.45] | 0.91 [0.79 to 0.98]
  Probability of decline: Week 145 | 0.22 [0.10 to 0.45] | 0.97 [0.87 to 1.00]
  Probability of decline: Week 193 | 0.26 [0.13 to 0.50] | 0.97 [0.87 to 1.00]
  Probability of decline: Week 241 | 0.40 [0.23 to 0.63] | 1.00 [0.87 to 1.00]
  Probability of decline: Week 289 | 0.54 [0.35 to 0.75] | 1.00 [0.87 to 1.00]
Statistical Analysis 1: Comparison: BMN 190-202 (300 mg) vs Natural History Comparator; Test type: Other; p < 0.0001, Cox Proportional Hazards model; Hazard Ratio (HR) = 0.14, 95% CI 2-sided [0.06 to 0.33]

2. Primary Outcome: Probability of Unreversed Motor-language (ML) Score of Zero.
Description: Motor and Language are each 0-3 point subscales in which 3 represents best function and 0 represents loss of function. Thus, the 0-6 point ML score was used as the primary mode of evaluation of loss of function.
  In 190-201, the primary endpoint was a responder endpoint: unreversed ML 2-point decline or score of 0 at Week 48 compared to the 50% rate expected in natural history using the 1-sample binomial test. For 190-202, the primary endpoint was revised to assess response over the full duration of follow-up. It is not clear, given the variable follow-up much greater than 48 weeks, what response rate is expected in natural history. For this reason, the assessment of the primary endpoint is based on comparing to natural history data and using the Kaplan-Meier method and Cox proportional hazards model with covariate adjustment (baseline ML score, age, genotype [common alleles], and sex).
Time Frame: Up to Week 289
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of decline
Groups:
- BMN 190-201/202 (300 mg): All study subjects administered BMN 190 300 mg by continuous Intracerebroventricular (ICV) infusion at a rate of 2.5 mL/hour for approximately 4 hours) every 14 days.
Arm/Group | BMN 190-201/202 (300 mg) | Natural History Comparator
Number analyzed (Participants) | 23 | 42
Probability of decline
  Probability of decline: Week 49 | 0.00 [0.00 to 0.00] | 0.03 [0.00 to 0.16]
  Probability of decline: Week 97 | 0.00 [0.00 to 0.00] | 0.38 [0.24 to 0.55]
  Probability of decline: Week 145 | 0.00 [0.00 to 0.00] | 0.78 [0.63 to 0.90]
  Probability of decline: Week 193 | 0.05 [0.01 to 0.28] | 0.94 [0.82 to 0.99]
  Probability of decline: Week 241 | 0.05 [0.01 to 0.28] | 0.97 [0.86 to 1.00]
  Probability of decline: Week 289 | 0.15 [0.05 to 0.39] | 1.00 [0.86 to 1.00]
Statistical Analysis 1: Comparison: BMN 190-201/202 (300 mg) vs Natural History Comparator; Test type: Other; p < 0.0001, Cox Proportional Hazards model; Hazard Ratio (HR) = 0.01

3. Secondary Outcome: Whole Brain Volume
Description: Percentage change from Baseline to Last Observation: Whole Brain volume
Time Frame: Baseline (Week 1 of BMN 190-201) to Week 289 / Last observation
Population: BMN 190-202: 24 subjects were enrolled in 190-201 at 5 clinic sites worldwide. One subject terminated from 190-201 after a single infusion and is not included in the Intent-to-Treat (ITT) population for 190-202. Study 190-202 final efficacy results include pooled data from the complete dataset from Study 190-201 & Study 190-202 for all subjects who received >1 dose (N=23).
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BMN 190-201/202 (300 mg)
Number analyzed (Participants) | 23
percentage change | -4.7 (10.54)

4. Secondary Outcome: Volume of Cerebrospinal Fluid
Description: Percentage Change from Baseline to last observation: Volume of cerebrospinal fluid
Time Frame: Baseline (Week 1 of BMN 190-201) to Week 289 / Last observation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BMN 190-201/202 (300 mg)
Number analyzed (Participants) | 23
percentage change | 8.5 (21.94)

5. Secondary Outcome: Volume of Total Cortical Gray Matter
Description: Percentage Change from Baseline to last observation: Volume of total cortical gray matter
Time Frame: Baseline (Week 1 of BMN 190-201) to Week 289 / Last observation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BMN 190-201/202 (300 mg)
Number analyzed (Participants) | 23
percentage change | -14.7 (10.25)

6. Secondary Outcome: Total White Matter Volume
Description: Percentage Change from Baseline to last observation: Total white matter volume
Time Frame: Baseline (Week 1 of BMN 190-201) to Week 289 / Last observation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BMN 190-201/202 (300 mg)
Number analyzed (Participants) | 23
percentage change | -2.4 (12.07)

7. Secondary Outcome: Whole Brain Apparent Diffusion Coefficient
Description: Change from Baseline to last observation Whole brain apparent diffusion coefficient
Time Frame: Baseline (Week 1 of BMN 190-201) to Week 289 / Last observation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm^2/s
Arm/Group | BMN 190-201/202 (300 mg)
Number analyzed (Participants) | 23
mm^2/s | 0.00 (0.030)

ADVERSE EVENTS:
Time Frame: Summaries of safety data were descriptive and designed to be inclusive of all adverse events reported in both the 190-201 and 190-202 studies. For each subject, adverse event (AE) data were collected from ICV access device implantation in Study 190-201, prior to any dose administration, to either 6 months after the last administration of study drug or the early termination visit in Study 190-202.
Description: 190-202 is the extension of treatment and follow-up for patients who enrolled in 190-201. Pooled data are presented since AE data for 190-202 were collected starting with ICV access device implantation in 190-201 (prior to any dose administration). Subjects who experienced more than 1 AE within a given MedDRA system organ class or preferred term were counted once within that system organ class or preferred term. Adverse events and deaths were not collected for Natural History participants.
Groups:
- BMN 190-202 (300 mg): Study 190-202 is the extension of treatment and follow-up for patients who enrolled in Study 190-201. Pooled data (Study 190-201/202; 24 subjects) are presented since adverse event data for Study 190-202 were collected starting with ICV access device implantation in Study 190-201 (prior to any dose administration).
Arm/Group | BMN 190-202 (300 mg)
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 21/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 190-202 (300 mg) (N=24)
Device related infection (Infections and infestations) | 7 (11)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Gastroenteritis (Infections and infestations) | 4 (4)
Pharyngitis bacterial (Infections and infestations) | 2 (3)
Pyelonephritis (Infections and infestations) | 2 (2)
Adenoviral upper respiratory infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (4)
Propionibacterium infection (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1)
Device end of service (Product Issues) | 13 (13)
Device leakage (Product Issues) | 1 (1)
Device malfunction (Product Issues) | 1 (1)
Pleocytosis (Nervous system disorders) | 3 (3)
Epilepsy (Nervous system disorders) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 7 (9)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Dental caries (Gastrointestinal disorders) | 2 (2)
Device deployment issue (Injury, poisoning and procedural complications) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Blindness (Eye disorders) | 1 (1)
CSF culture positive (Investigations) | 1 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 190-202 (300 mg) (N=24)
Hypotension (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 3 (3)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Hypersensitivity (Immune system disorders) | 10 (16)
Seasonal allergy (Immune system disorders) | 3 (4)
Pyrexia (General disorders) | 20 (219)
Gait disturbance (General disorders) | 12 (15)
Abasia (General disorders) | 3 (3)
Complication associated with device (General disorders) | 3 (3)
Developmental delay (General disorders) | 3 (3)
Pain (General disorders) | 3 (4)
Feeling jittery (General disorders) | 2 (5)
Sleep disorder (Psychiatric disorders) | 9 (14)
Insomnia (Psychiatric disorders) | 5 (5)
Irritability (Psychiatric disorders) | 5 (6)
Agitation (Psychiatric disorders) | 4 (5)
Abnormal behaviour (Psychiatric disorders) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 8 (36)
Contusion (Injury, poisoning and procedural complications) | 8 (11)
Head injury (Injury, poisoning and procedural complications) | 3 (8)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Device deployment issue (Injury, poisoning and procedural complications) | 2 (2)
Device difficult to use (Injury, poisoning and procedural complications) | 2 (7)
Laceration (Injury, poisoning and procedural complications) | 2 (6)
Limb injury (Injury, poisoning and procedural complications) | 2 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2)
Procedural vomiting (Injury, poisoning and procedural complications) | 2 (2)
Stoma site reaction (Injury, poisoning and procedural complications) | 2 (3)
Body temperature increased (Investigations) | 4 (5)
CSF red blood cell count positive (Investigations) | 3 (3)
Oxygen saturation decreased (Investigations) | 3 (11)
CSF test abnormal (Investigations) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7)
Anaemia (Blood and lymphatic system disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 16 (250)
Seizure (Nervous system disorders) | 14 (201)
Epilepsy (Nervous system disorders) | 13 (180)
Tremor (Nervous system disorders) | 11 (13)
Extensor plantar response (Nervous system disorders) | 9 (13)
Myoclonus (Nervous system disorders) | 10 (24)
Petit mal epilepsy (Nervous system disorders) | 8 (22)
Partial seizures (Nervous system disorders) | 7 (15)
Pleocytosis (Nervous system disorders) | 6 (6)
Speech disorder (Nervous system disorders) | 6 (6)
Language disorder (Nervous system disorders) | 5 (5)
Dyskinesia (Nervous system disorders) | 4 (11)
Athetosis (Nervous system disorders) | 4 (6)
Headache (Nervous system disorders) | 4 (13)
Ataxia (Nervous system disorders) | 3 (3)
Atonic seizures (Nervous system disorders) | 3 (6)
Myoclonic epilepsy (Nervous system disorders) | 3 (6)
Muscle spasticity (Nervous system disorders) | 3 (3)
Movement disorder (Nervous system disorders) | 3 (3)
Seizure cluster (Nervous system disorders) | 3 (7)
Clonus (Nervous system disorders) | 2 (2)
Chorea (Nervous system disorders) | 2 (2)
Balance disorder (Nervous system disorders) | 2 (2)
Drop attacks (Nervous system disorders) | 2 (2)
Hypotonia (Nervous system disorders) | 2 (2)
Status epilepticus (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (4)
Dystonia (Nervous system disorders) | 3 (3)
Visual impairment (Eye disorders) | 11 (16)
Blindness (Eye disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 13 (22)
Vomiting (Gastrointestinal disorders) | 19 (78)
Dysphagia (Gastrointestinal disorders) | 13 (26)
Dental caries (Gastrointestinal disorders) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 6 (10)
Diarrhoea (Gastrointestinal disorders) | 9 (19)
Salivary hypersecretion (Gastrointestinal disorders) | 3 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 3 (4)
Teething (Gastrointestinal disorders) | 3 (3)
Oesophagitis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Device end of service (Product Issues) | 13 (13)
Device leakage (Product Issues) | 4 (10)
Needle issue (Product Issues) | 9 (11)
Device malfunction (Product Issues) | 4 (9)
Device issue (Product Issues) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 3 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (5)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 21 (73)
Gastroenteritis (Infections and infestations) | 9 (15)
Device related infection (Infections and infestations) | 9 (14)
Viral upper respiratory tract infection (Infections and infestations) | 19 (46)
Rhinitis (Infections and infestations) | 13 (22)
Conjunctivitis (Infections and infestations) | 6 (7)
Viral infection (Infections and infestations) | 9 (16)
Pharyngitis (Infections and infestations) | 7 (14)
Respiratory tract infection (Infections and infestations) | 6 (9)
Influenza (Infections and infestations) | 5 (5)
Rhinovirus infection (Infections and infestations) | 4 (8)
Bronchitis (Infections and infestations) | 3 (4)
Lower respiratory tract infection (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 3 (8)
Corona virus infection (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 2 (2)
Oral herpes (Infections and infestations) | 2 (7)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Epstein-Barr virus infection (Infections and infestations) | 2 (4)
Pharyngitis bacterial (Infections and infestations) | 2 (3)
Pneumonia (Infections and infestations) | 2 (5)
Tonsillitis bacterial (Infections and infestations) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 2 (2)
Varicella (Infections and infestations) | 2 (2)
Pyelonephritis (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 5 (12)
Otitis media (Infections and infestations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restrictions on the PI are that (i) they cannot publish results communications until after the multicenter dataset is published, (ii) the sponsor has an opportunity to review results communications prior to public release, and (iii) the sponsor can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days.

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT02485899/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT02485899/SAP_001.pdf